CLINICAL TRIAL: NCT04286620
Title: ASSESSMENT OF INTRA-OPERATIVE AND EARLY POST-OPERATIVE LASIK COMPLICATIONS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed saad, House officer, Assiut University
Other Study IDs: LASIK complications
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Cornea
Keywords: LASIK complications
MeSH Terms: conditions — Corneal Diseases | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LASIK — Correcting errors of refraction

SUMMARY:
To discuss the prevalence of intra-operative and early post-operative complications of LASIK among individuals who underwent LASIK procedure and review the symptoms, findings, and management options.

DETAILED DESCRIPTION:
In recent years, a number of possible surgical procedures in ophthalmology has offered patients an alternative to spectacles or contact lenses. Several laser and non-laser refractive surgical procedures have been used to modify the shape of the cornea and correct myopia, hyperopia, astigmatism, and presbyopia. Introduction of the excimer laser to reshape the cornea has resulted in remarkable developments in the correction of refractive errors. Combined with other advanced ophthalmic instruments, laser refractive eye surgery has resulted in a substantial increase in the safety, efficacy, and predictability of surgical outcomes.

Refractive surgery has enabled individuals to enter occupations they were previously precluded from due to their vision.Laser in situ keratomileusis (LASIK) surgery is one of the most common surgeries performed worldwide to correct refractive errors and reduce dependence on eyeglasses or contact lenses. In addition, patient satisfaction following LASIK is commonly reported as high and studies of the visual and refractive outcome of LASIK for the treatment of myopia and astigmatism have reported great success.

LASIK, compared to photorefractive keratectomy (PRK), has low postoperative discomfort, early visual rehabilitation and decreased postoperative haze. LASIK involves an additional procedure of creating a corneal flap. This may result in complications related to the flap, interface and underlying stromal bed. The common flap-related complications include thin flap, button holing, free caps, flap dislocation, torn flap, incomplete cut, and flap striae. The interface complications of diffuse lamellar keratitis, epithelial ingrowth and microbial keratitis are potentially sight threatening. After LASIK, there is a long period of sensory denervation leading to the complication of dry eyes. The refractive complications include under-correction, over-correction, regression, irregular astigmatism, and visual aberrations.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are scheduled for LASIK surgery

Exclusion Criteria:

* history of previous ocular surgery, and inadequate follow up.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Parameters to be included: demographic data, history, symptoms, post-operative uncorrected and best corrected visual acuities, examination findings, and treatment recommendations.
  Documentation of complications.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of Intra-operative and early post-operative complications of LASIK | Baseline
  Assessment of post-LASIK complications

CONTACTS AND LOCATIONS:
Overall Officials: Tarek A Mohamed, Professor, Study Director — Ophthalmology department, faculty of medicine, Assiut university hospital; Dalia M El-Sebity, Ass.prof., Study Director — Ophthalmology department, faculty of medicine, Assiut university hospital; Khaled A Mohammed, Ass.prof., Study Director — Ophthalmology department, faculty of medicine, Assiut university hospital